CLINICAL TRIAL: NCT00969020
Title: The Effect of Remote Rehabilitation Support Via a Telemedicine Solution for Patients Undergoing an Optimized Fast-track Orthopedic Surgery Procedure With the Implementation of a Total Hip Arthroplasty.
Brief Title: A Telemedicine Solution for Remote Support of Rehabilitation, for Patients Undergoing, Total Hip Arthroplasty Surgery
Acronym: RRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Collaborators: Caretech Innovation (Unknown); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Martin Vesterby, MD, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009-RSI-RRS
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Quality of Life; Anxiety
Keywords: Length of stay; Timed up and go
MeSH Terms: conditions — Anxiety Disorders | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Active Comparator): RRS via telemedicine. By developing the concept of Remote Rehabilitation Support (RRS) the investigators will try to bring preoperative education of the patient, dissemination of information and postoperative support to a new level.
  Interventions: Procedure: remote rehabilitation support
- Standard (No Intervention): The standard procedure for THA used under The Lundbeck Center for fast track hip and knee surgery

INTERVENTIONS:
Procedure: remote rehabilitation support — An information technology solution containing RRS. The way it supports,, informs and educates the patient and support person, provides an opportunity for communication between the patient and the surgeons, physiotherapists and nurses at the hospital.
  Other Names: Rehabilitation; Fast-track
  Arms: Telemedicine

SUMMARY:
The RRS project is a Randomized Clinical Trial documenting the effect of Remote Rehabilitation and Support via a telemedicine solution for patients undergoing an optimized fast-track orthopedic surgery procedure with the implementation of a total hip arthroplasty. With the telemedicine solution the investigators will support and try to motivate the patient to be discharged after only one day of hospitalization.

DETAILED DESCRIPTION:
This PhD study evaluates the effect of an information technology solution containing RRS. The way it supports, informs and educates the patient and support person, provides an opportunity for communication between the patient and the surgeons, physiotherapists and nurses at the hospital.

The parameters evaluated will be: Length of stay, health-related quality-of-life (HRQOL), functional outcome, pain, anxiety, complications and an evaluation of the socio-economic effect.

The aim of the study generates the following hypotheses and focus for publication

* Length of stay is lower for the intervention group compared to the control group.
* The average quality of life measured with EQ-5D will either be the same or higher when comparing the intervention group with the control group.
* Compared to the control group the functional outcome of the intervention group measured with Oxford Hip Score (OHS) and Timed Up and Go (TUG) will be the same or better.
* Complications measured as luxations, infections, and reoperations are the same or lower in the intervention group compared to the control group.
* There will be a correlation between patients with the highest level of psychological problems and symptoms of psychopathology measured with Symptom Checklist-90-R, and the postoperative outcome measured with EQ5D, anxiety and TUG.
* There will be a correlation between support persons with the highest level of psychological problems and symptoms of psychopathology measured with Symptom Checklist-90-R, and the postoperative outcome measured with EQ5D, anxiety and TUG for the patient they are related to.
* The socio-economic costs will be lower for the intervention group compared to the control group based on self reported data and data collected from official databases. This study will be conducted as a piggy back to the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified to go trough at joint-care procedure after the guidelines from Regionshospitalet Silkeborg.

Exclusion Criteria:

* Previous hip surgery with the implantation of a total hip arthroplasty.
* Patients living more than approximately 60 kilometers from the Regionshospitalet Silkeborg.
* Patients with no 3G tele-net at their home address.
* Patients with the need of Danish interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
EQ5D | 12 months
LOS | up to 5 days
  Length of Stay

SECONDARY OUTCOMES:
SCL-90-r | day 0
  psychological problems and symptoms of psychopathology
TUG | day 90
  Time up and go
anxiety | Day 90
  VAS - anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Professor, Study Director — University of Aarhus, Orthopaedic surgical research
Locations (1):
- Regionshospitalet SIlkeborg, Silkeborg, Silkeborg, Denmark